CLINICAL TRIAL: NCT03572530
Title: Infusion of 5-Azacytidine (5-AZA) Into the Fourth Ventricle or Resection Cavity in Children and Adults With Recurrent Posterior Fossa Ependymoma: A Phase I Study
Brief Title: Infusion of 5-Azacytidine (5-AZA) Into the Fourth Ventricle in Patients With Recurrent Posterior Fossa Ependymoma
Acronym: 5-AZA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, David Ilan Sandberg, Professor, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-18-0309
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Recurrent Ependymoma
MeSH Terms: conditions — Ependymoma | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- group 1 (Experimental): 5-Azacytidine (5-AZA) group 1: Enrolled patients will undergo surgical placement of a ventricular catheter into the fourth ventricle that will be attached to a subcutaneously placed reservoir. Patients will be divided into 3 dose groups and receive 8 weeks of intraventricular 5-AZA (12 mg) into the fourth ventricle. Patients in Group 1 will receive two 5-AZA infusions every week.
  Interventions: Drug: 5-Azacytidine (5-AZA) group 1
- group 2 (Experimental): 5-Azacytidine (5-AZA) group 2: Enrolled patients will undergo surgical placement of a ventricular catheter into the fourth ventricle that will be attached to a subcutaneously placed reservoir. Patients will be divided into 3 dose groups and receive 8 weeks of intraventricular 5-AZA (12 mg) into the fourth ventricle. Patients in Group 2 will receive three 5-AZA infusions every week.
  Interventions: Drug: 5-Azacytidine (5-AZA) group 2
- group 3 (Experimental): 5-Azacytidine (5-AZA) group 3: Enrolled patients will undergo surgical placement of a ventricular catheter into the fourth ventricle that will be attached to a subcutaneously placed reservoir. Patients will be divided into 3 dose groups and receive 8 weeks of intraventricular 5-AZA (12 mg) into the fourth ventricle. Patients in Group 3 will receive four 5-AZA infusions every week.
  Interventions: Drug: 5-Azacytidine (5-AZA) group 3

INTERVENTIONS:
Drug: 5-Azacytidine (5-AZA) group 1 — 5-AZA (12 mg) will be prepared in preservative-free normal saline to a total volume of 1.2ml. 5-AZA will be infused over a minimum of 30 seconds. 5-AZA will be followed by a 1 ml preservative-free normal saline flush over a minimum of 30 seconds.
  Patients will receive two, three, or four 5-AZA infusions per week depending on the dosing algorithm (see below). We refer to these dosing schedules as dose 1, 2, or 3.
  Patients assigned to dose 1 will receive two 5-AZA infusions per week (typically Monday and Thursday but may be given on other days based upon logistical considerations) for 8 consecutive weeks.
  Other Names: Vidaza
  Arms: group 1
Drug: 5-Azacytidine (5-AZA) group 2 — 5-AZA (12 mg) will be prepared in preservative-free normal saline to a total volume of 1.2ml. 5-AZA will be infused over a minimum of 30 seconds. 5-AZA will be followed by a 1 ml preservative-free normal saline flush over a minimum of 30 seconds.
  Patients will receive two, three, or four 5-AZA infusions per week depending on the dosing algorithm (see below). We refer to these dosing schedules as dose 1, 2, or 3.
  Patients assigned to dose 2 will receive three 5-AZA infusions per week (typically Monday, Wednesday, and Friday but may be given on other days based upon logistical considerations) for 8 consecutive weeks.
  Other Names: Vidaza
  Arms: group 2
Drug: 5-Azacytidine (5-AZA) group 3 — 5-AZA (12 mg) will be prepared in preservative-free normal saline to a total volume of 1.2ml. 5-AZA will be infused over a minimum of 30 seconds. 5-AZA will be followed by a 1 ml preservative-free normal saline flush over a minimum of 30 seconds.
  Patients will receive two, three, or four 5-AZA infusions per week depending on the dosing algorithm (see below). We refer to these dosing schedules as dose 1, 2, or 3.
  Patients assigned to dose 3 will receive four 5-AZA infusions per week (on any 4 weekdays based upon logistical considerations) for 8 consecutive weeks.
  Other Names: Vidaza
  Arms: group 3

SUMMARY:
This study seeks to determine the optimum dose frequency of 5-Azacytidin (5-AZA) infusions into the fourth ventricle of the brain. The study's primary objective is to establish the maximum tolerated dose for infusions of 5-Azacytidine into the fourth ventricle in patients with recurrent ependymoma. The study's secondary objective is to assess the antitumor activity of 5-Azacytidine infusions into the fourth ventricle based upon imaging studies and cytology.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Patients with histologically verified ependymoma, with recurrence or progression anywhere in the brain and/or spine. Patients are also eligible if they have refractory disease, which will be defined as residual tumor which has not been completely cleared despite prior treatments. To be eligible, patients' disease must have originated in the posterior fossa of the brain
* Patient must have either measurable or evaluable tumor as assessed by MRI of the brain and total spine
* An implanted catheter in the fourth ventricle or posterior fossa tumor cavity attached to a ventricular access device or agreement to have one placed.
* A minimum of 7 days between last dose of systemic chemotherapy and/or radiation therapy and first infusion of 5-AZA into fourth ventricle
* Life expectancy of at least 12 weeks in the opinion of the principal investigator
* Lansky score of 50 or greater if ≤16 years of age or Karnofsky score of 50 or greater if > 16 years of age
* Existing neurological deficits must have been stable for a minimum of 1 week prior to study enrollment
* Patients must have recovered from the acute toxic effects of all prior anticancer chemotherapy
* Adequate bone marrow function defined by peripheral absolute neutrophil count (ANC) ≥ 500/μL, platelet count ≥ 50,000/μL (transfusion independent), and hemoglobin ≥ 9.0 gm/dL (may receive RBC transfusions)
* Patient or patient's legal representative, parent(s), or guardian able to provide written informed consent.

Exclusion Criteria:

* Enrolled in another treatment protocol
* Has received another investigational or chemotherapy agent or radiation therapy within 7 days prior to 5-AZA infusion into the fourth ventricle
* Evidence of untreated infection
* Pregnant or lactating women

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-24 (Actual)

PRIMARY OUTCOMES:
Number of participants who experienced dose-limiting toxicity (DLT) | 8 weeks
  Dose-limiting toxicity will be defined as any of the following events:
  New neurological deficit (grade 3 or higher) probably or definitely attributed to intraventricular 5-azacytidine infusions.
  New adverse event involving any organ probably or definitely attributed to intraventricular 5-azacytidine infusions with the specific exclusion of: Grade 3 or higher nausea and vomiting < 3 days duration and grade 3 or higher headache < 3 days duration.

SECONDARY OUTCOMES:
Number of participants with disease progression as assessed by magnetic resonance imaging (MRI) | 1 day after surgery to remove tumor (which is about 1 week before the first infusion)
  The PI and radiologist will determine Response to treatment according to the following three categories. Disease progression corresponds with the "Progressive Disease" category.
  Complete Response (CR): Disappearance of all non-target lesions. Stable Disease (SD) / Incomplete Response (IR): The persistence of one or more non-target lesions.
  Progressive Disease (PD): The appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Number of participants with disease progression as assessed by magnetic resonance imaging (MRI) | 8 weeks after first infusion
  The PI and radiologist will determine Response to treatment according to the following three categories. Disease progression corresponds with the "Progressive Disease" category.
  Complete Response (CR): Disappearance of all non-target lesions. Stable Disease (SD) / Incomplete Response (IR): The persistence of one or more non-target lesions.
  Progressive Disease (PD): The appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.

CONTACTS AND LOCATIONS:
Overall Officials: David I Sandberg, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lang F, Liu Y, Chou FJ, Yang C. Genotoxic therapy and resistance mechanism in gliomas. Pharmacol Ther. 2021 Dec;228:107922. doi: 10.1016/j.pharmthera.2021.107922. Epub 2021 Jun 23. PMID 34171339